CLINICAL TRIAL: NCT01107093
Title: A Prospective, Randomized, Double-blind, Cross-Over Study to Compare the Capacity to Prevent Follicular Rupture of CDB-2914 With Placebo, When Administered After the Ovulatory Process Has Been Triggered by the LH Surge
Brief Title: Comparison of CDB-2914 Versus Placebo in the Prevention of Follicular Rupture Post-luteinizing Hormone (LH) Surge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Erin Gainer, R&D Director, HRA Pharma
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2914-007
Record Dates: First submitted 2010-04-12; First posted 2010-04-20 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Contraception
MeSH Terms: interventions — ulipristal; ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CDB-2914 (Active Comparator)
  Interventions: Drug: CDB-2914 (ulipristal acetate)

INTERVENTIONS:
Drug: CDB-2914 (ulipristal acetate) — single oral dose of 30 mg
  Arms: CDB-2914
Drug: Placebo — single oral dose
  Arms: Placebo

SUMMARY:
Evaluation of the effect of a single dose of CDB-2914, as compared to placebo, administered after the onset of the LH surge on the outcome of the leading ovary follicle:

* echographic follicle rupture
* inhibition of follicle rupture
* luteal phase progesterone levels
* anovulatory progesterone levels

ELIGIBILITY:
Inclusion Criteria:

* Women of good general health aged 18 - 35 years
* Not at risk of pregnancy
* Regular menstrual cycles of 24-35 days duration
* Not pregnant
* Intact uterus and ovaries
* Haemoglobin ≥ 11 g/dl
* Normal laboratory tests and normal TSH
* Willing to abstain from any use of hormonal contraception until study completion
* No current use of hormonal contraception and having had at least one complete menstrual cycle (2 menses) since termination of previous hormonal contraception
* Had at least one complete menstrual cycle (2 menses) following delivery, miscarriage or induced abortion
* Able to give voluntary, written informed consent, and agreeing to observe all study requirements for 5 complete menstrual cycles

Exclusion Criteria:

* Current participation in any other trial of an investigational medicine
* Known hypersensitivity to the ingredients of the test active substances or excipients
* Suspected hyperplasia or carcinoma of the endometrium
* Current pregnancy as confirmed by positive serum beta-hCG at screening
* Desire to get pregnant before the planned end of the study participation
* Currently breastfeeding
* Abnormal Pap smear
* Cancer (past history of any carcinoma or sarcoma)
* Known or suspected alcoholism or drug abuse
* Abnormal thyroid status
* Body mass index > 32
* Current use of hormonal contraception
* Use of hormonal emergency contraception since last menstrual period
* Severe asthma insufficiently controlled by oral glucocorticoids
* Hereditary galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Inhibition of follicular rupture | within 6 days after treatment intake
  Inhibition is calculated as the number of subjects exhibiting no dominant follicle rupture, divided by the total number of subjects having received treatment

SECONDARY OUTCOMES:
Appearance or absence of a corpus luteum | during the 6 days following treatment intake
Growth pattern of leading follicle
  number of cycles exhibiting atresia (diameter decrease ≥25%), or continued growth (diameter increase ≥25%), or interrupted growth (size remains within ±25% of the follicle size at the time of treatment)
Presence or absence of a surge of serum luteinizing hormone (LH) levels
  The onset of an LH surge is defined as the occurrence of the first single serum LH value whose level is at least 50% higher than the mean of the last two previous measurements, or higher than the last previous measurement if only one previous LH level is available.
Menstrual cycle length in comparison to the subject's reported baseline average cycle length and to her placebo-treated cycle length
Incidence of intermenstrual bleeding and treatment-emergent adverse events
Incidence of adverse events and occurrence of abnormal laboratory safety variables in comparison with baseline
Incidence of ovarian cysts after CDB-2914 treatment

CONTACTS AND LOCATIONS:
Locations (2):
- ICMER, Santiago, Chile
- Clinica de PROFAMILIA, Santo Domingo, Dominican Republic

REFERENCES:
- [Result] Brache V, Cochon L, Jesam C, Maldonado R, Salvatierra AM, Levy DP, Gainer E, Croxatto HB. Immediate pre-ovulatory administration of 30 mg ulipristal acetate significantly delays follicular rupture. Hum Reprod. 2010 Sep;25(9):2256-63. doi: 10.1093/humrep/deq157. Epub 2010 Jul 15. PMID 20634186